CLINICAL TRIAL: NCT03026348
Title: Safety and Immunogenicity Study to Evaluate Single- or Two-Dose Regimens Of RSV F Vaccine With and Without Aluminum Phosphate or Matrix-M1™ Adjuvants In Clinically-Stable Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RSV-E-205
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Respiratory Syncytial Viruses
Keywords: RSV
MeSH Terms: interventions — Matrix-M

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- Treatment Group A (Active Comparator): Day 0 RSV F Vaccine 135µg/0.5mL Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine; Other: Phosphate Buffer
- Treatment Group B (Active Comparator): Day 0 Treatment / Formulation 1 Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine with Aluminum Phosphate Adjuvant; Other: Phosphate Buffer
- Treatment Group C (Active Comparator): Day 0 Treatment / Formulation 1 Day 21 Treatment / Formulation 1
  Interventions: Biological: RSV F Vaccine with Aluminum Phosphate Adjuvant
- Treatment Group D (Active Comparator): Day 0 Treatment / Formulation 2 Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine with Aluminum Phosphate Adjuvant; Other: Phosphate Buffer
- Treatment Group E (Active Comparator): Day 0 Treatment / Formulation 2 Day 21 Treatment / Formulation 2
  Interventions: Biological: RSV F Vaccine with Aluminum Phosphate Adjuvant
- Treatment Group F (Active Comparator): Day 0 Treatment / Formulation 3 Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant; Other: Phosphate Buffer
- Treatment Group G (Active Comparator): Day 0 Treatment / Formulation 3 Day 21 Treatment / Formulation 3
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant
- Treatment Group H (Active Comparator): Day 0 Treatment / Formulation 4 Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant; Other: Phosphate Buffer
- Treatment Group J (Active Comparator): Day 0 Treatment / Formulation 4 Day 21 Treatment / Formulation 4
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant
- Treatment Group K (Active Comparator): Day 0 Treatment / Formulation 5 Day 21 Phosphate Buffer
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant; Other: Phosphate Buffer
- Treatment Group L (Active Comparator): Day 0 Treatment / Formulation 5 Day 21 Treatment / Formulation 5
  Interventions: Biological: RSV F Vaccine; Biological: Matrix-M1 Adjuvant
- Treatment Group M (Placebo Comparator): Day 0 Phosphate Buffer Day 21 Phosphate Buffer
  Interventions: Other: Phosphate Buffer

INTERVENTIONS:
Biological: RSV F Vaccine with Aluminum Phosphate Adjuvant
  Arms: Treatment Group B; Treatment Group C; Treatment Group D; Treatment Group E
Biological: RSV F Vaccine
  Arms: Treatment Group A; Treatment Group F; Treatment Group G; Treatment Group H; Treatment Group J; Treatment Group K; Treatment Group L
Biological: Matrix-M1 Adjuvant
  Arms: Treatment Group F; Treatment Group G; Treatment Group H; Treatment Group J; Treatment Group K; Treatment Group L
Other: Phosphate Buffer
  Arms: Treatment Group A; Treatment Group B; Treatment Group D; Treatment Group F; Treatment Group H; Treatment Group K; Treatment Group M

SUMMARY:
This is a randomized, observer-blind, trial in clinically-stable older adults. Up to 300 eligible older adults 60 through 80 years of age will be enrolled at a 1:1 ratio into multiple dose/formulation treatment arms. Safety and immunogenicity data through Day 56 will be used to select a vaccine candidate to potentially evaluate in a Part 2 study. Proportions of subjects in various strata will not be pre-specified and the goal will be to achieve an approximately equal distribution of subjects with these characteristics across the treatment groups. Serology measures consistent with the study outcomes will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 60 through 80 years of age who are ambulatory and live in the community or in an assisted-living facility that provides minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living. Subjects may have one or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Absence of changes in medical therapy within one month due to treatment failure or toxicity (dose adjustments of ongoing therapies for optimal effect, or replacements within a class of drugs due to convenience or cost, will be deemed acceptable),
   * Absence of medical events qualifying as SAEs within one month of the planned vaccination on Day 0, and
   * Absence of known, current, and life-limiting diagnoses which, in the opinion of the investigator, render survival to completion of the protocol unlikely.
2. Willing and able (on both a physical and cognitive basis) to give informed consent prior to study enrollment. To complete the consent process, all qualifying subjects will correctly answer at least 4 out of 5 questions of the informed consent form (ICF) comprehension assessment in no more than 2 attempts.
3. Able to comply with study requirements. As the protocol procedures involve telephone contacts for safety ascertainment, eligible subjects must have a reliable access to a telephone.

Exclusion Criteria:

1. Received any prior RSV vaccine.
2. Participation in research involving any additional investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
3. History of a serious reaction to any prior vaccination or a history of Guillain-Barré syndrome (GBS) within 6 weeks of any prior influenza immunization.
4. Receipt of inactivated influenza vaccine within 14 days prior to the Day 0 dose of test article or any other vaccine within the 4 weeks prior to the Day 0 dose of test article.
5. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
6. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
7. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
8. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C on the planned day of vaccine administration).
9. Known disturbance of coagulation. Potential subjects receiving aspirin, clopidogrel, prasugrel, dipyridamole, dabigatran, apixaban, rivaroxaban, or warfarin under good control for cardiovascular prophylaxis or prophylaxis of thromboembolic disease or stroke in the setting of atrial fibrillation will NOT be excluded.
10. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
11. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic, cognitive, or psychiatric conditions deemed likely to impair the quality of study compliance or safety reporting).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01; Primary Completion 2017-04 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibody titers to at least one RSV/A strain | Day 0, 21, 28
Subjects with solicited local and systemic AEs occurring within the 7-day period following dosings on Day 0 and Day 21 and all adverse events, solicited and unsolicited, occurring within the 56-day period of Day 0. | Day 0 - Day 6, Day 21 - Day 27; Day 0 - Day 56

SECONDARY OUTCOMES:
Serum concentrations of antibodies competitive with palivizumab (i.e., PCA) for binding to the RSV F protein. | Day 0, 21, 28, 56, 119, 385
Serum IgG antibody concentrations as ELISA units (EUs) specific for the F protein antigen. | Day 0, 21, 28, 56, 119, 385
Counts of IFN-γ spot forming units following in vitro stimulation of Day 0, Day 7, and Day 28 PBMC isolates with RSV F peptides. | Day 0, 7, 28
Counts and proportions of Day 0, Day 7, and Day 28 peripheral blood T cells positive by intracellular staining for IL-2, IFN-γ, or TNF-α production (alone or any combination thereof) following in vitro stimulation with RSV F peptides. | Day 0, 7, 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (5):
- Australia (5):
  - Research Site AU004, Sydney, New South Wales
  - Research Site AU005, Herston, Queensland
  - Research Site AU002, Adelaide, South Australia
  - Research Site AU006, Prahran, Victoria
  - Resarch Site AU001, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided